CLINICAL TRIAL: NCT06562205
Title: External Evaluation of PAP Systems: Comparison of PAP Flow Generators Machines, Mask Systems and Tubing
Brief Title: PAP Systems External Clinical Studies (ECS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SLP-24-08-01
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: his is an open label, prospective, randomized cross over (or single arm) study designed to support the development of new accessories for PAP devices.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAP System A (with Amalfi) then PAP System B (with CLA11) (Experimental): Participants will be asked to take home the investigational PAP system (Amalfi) to use at night while they sleep in place of their own PAP system. The participant's therapy and comfort settings will not be altered. Participants will be randomized as to the order they will trial PAP System A and PAP System B. This arm will first use the Amalfi for 7 days and then use the CLA 11 for 7 days.
  Interventions: Device: PAP System A (with Amalfi) then PAP System B (with CLA11); Device: PAP System B (with CLA11) then PAP System A (with Amalfi)
- PAP System B (with CLA11) then PAP System A (with Amalfi) (Active Comparator): Participants will be asked to take home the comparator PAP system B (CLA 11) to use at night while they sleep in place of their own PAP system. The participant's therapy and comfort settings will not be altered. Participants will be randomized as to the order they will trial PAP System B and PAP System A. This arm will first use the CLA 11 for 7 days and then use the Amalfi for 7 days.
  Interventions: Device: PAP System A (with Amalfi) then PAP System B (with CLA11); Device: PAP System B (with CLA11) then PAP System A (with Amalfi)

INTERVENTIONS:
Device: PAP System A (with Amalfi) then PAP System B (with CLA11) — PAP System A (with Amalfi) for 7 days followed by PAP System B (with CLA11) for 7 days
Device: PAP System B (with CLA11) then PAP System A (with Amalfi) — PAP System B (with CLA11) for 7 days followed by PAP System A (with Amalfi) for 7 days

SUMMARY:
This is a pre-market study for ongoing product development aiming to explore the usability and performance of the study PAP systems.

DETAILED DESCRIPTION:
This is an open label, prospective, randomized cross over (or single arm) study for ongoing product development of new accessories for PAP devices. This generic protocol provides a framework methodology for how these ongoing studies will be conducted. This protocol then is used in a number of smaller sub-studies phases, each of which will have their own sub-protocol outlining the exact specifics of the study.

The studies could be run face-to-face or remotely.

Participants who met the inclusion/exclusion criteria will be contacted. Recruitment will be done via emails. Participants will be explained the details of the trial and those who wish to take part will be invited to a selected site for the first study visit.

Visit 1: Participants will provide written informed consent. Participants will be shown the PAP systems and trial them for fit and comfort. Participants may be asked initial questions on their first thoughts on the PAP systems. If the participant and assessor are happy to proceed, the participants will use the loan PAP system for trial.

Visit 2: After trialing the PAP systems, participants will be asked to complete a questionnaire regarding the appeal, comfort, and usability of the PAP system(s). Depending on sub-study protocol, participants will then take the second PAP system home to test.

Visit 3: The participant will return the loan PAP system to the assessor. The participants' questionnaire responses will be reviewed. This concludes the participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who ≥ 18 years of age
* Participants being treated for OSA for ≥ 3 months
* Participants currently using a suitable PAP system(s)
* Participants who can trial the PAP systems for up to 7 nights each

Additional criteria for remote studies:

* Participants currently using PAP device compatible with AirView, or with download capacity from PAP machine from data cards
* Participants who have access to video call equipment

Exclusion Criteria:

* Participants using Bilevel flow generators
* Participants who are or may be pregnant
* Participants with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Participants believed to be unsuitable for inclusion by the researcher
* Participants who or whose bed partner has implantable medical devices which may contraindicate against masks with magnetic clips (exclusion criteria for study masks with magnetic clips only)
* Participants who are currently enrolled in other clinical studies

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
(usability) Comparison of the usability of an investigational component/s of the PAP system to a comparison component/s of the PAP system and/or Criterion Score of 6 | 6 weeks
  Hypothesis: The investigational component/s of the PAP system will be equivalent to the comparison component/s of the PAP system and/or Criterion Score of 6
  Subjective usability scores will be collected from participants on each usability item (e.g., comfort, seal, ease of use). Scores will be collected using an 11-point Likert Scale where a score of 10 is considered very favorable, and a score of 0 is very unfavorable
(efficacy) Comparison of the investigational component/s of the PAP system efficacy (AHI) to a comparison component/s of the PAP system and/or clinically relevant data | 6 weeks
  Hypothesis: The investigational component/s of the PAP system will be equivalent to the comparison component/s of the PAP system and/or clinically relevant data
  Objective data stored in the CPAP device will be downloaded wirelessly using a computer program (AirView or ResScan, ResMed). An Apnea hypopnea index (AHI) automatically analyzed by the program will be used. Typically, an AHI <5 demonstrates efficacious treatment.

IPD SHARING:
Plan to Share IPD: No